CLINICAL TRIAL: NCT07313124
Title: The Efficiency and Safety of Single Drug Versus Combinations of Antihyperlipidemic Agents in Treatment of Cardiovascular Diseases
Brief Title: Comparative Study Between Antihyperlipidemic Agents in Treatment of Cardiovascular Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Lecturer of Clinical Pharmacy, Beni-Suef University, Egypt, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/05012025/Elsaid
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases (CVD)
Keywords: Antihyperlipidemic; Cardiovascular diseases; Rosuvastatin
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RosUvastatin (Experimental): Patients will receive to rosuvastatin 20 mg
  Interventions: Drug: rosuvastatin drug
- rosuvastatin ezetimibe10/10mg. (Active Comparator): Patients will receive rosuvastatin ezetimibe10/10mg.
  Interventions: Combination Product: Patients received rosuvastatin ezetimibe10/10mg

INTERVENTIONS:
Drug: rosuvastatin drug — Patients randomized to receive rosuvastatin 20 mg
  Arms: RosUvastatin
Combination Product: Patients received rosuvastatin ezetimibe10/10mg — Patients received rosuvastatin ezetimibe10/10mg
  Arms: rosuvastatin ezetimibe10/10mg.

SUMMARY:
The goal of this clinical trial is to study the efficiency and safety of using combinations of antihyperlipidemic agents with a single drug to treat cardiovascular diseases.

The main questions it aims to answer are:

* Which approach is more effective rosuvastatin monotherapy or rosuvastatin ezetimibe combination antihyperlipidemic for patients with cardiovascular diseases (CVDs)?
* What medical problems do participants could when taking antihyperlipidemic drugs? Researchers will compare rosuvastatin 20 mg or rosuvastatin ezetimibe10/10mg to see the effectiveness and safety of these drugs in patients with CVDs.

Participants will:

* Patients will randomize to either rosuvastatin 20 mg or rosuvastatin ezetimibe10/10mg.
* Patients will be followed up to 12 weeks after starting treatment.
* All the patients will be subjected to: Full sheet taking, including detailed history and diagnosis of the case, Baseline Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) tests& after 24 weeks of treatment, Lipid Profile, creatine kinase (CK) test, Creatine kinase-MB (CK-MB) test.

ELIGIBILITY:
Inclusion Criteria:

Adults above 18 years, Dyslipidemic patients

Exclusion Criteria:

Young people under 18 years old pregnant women lactating women Children Hypersensitivity Renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Creatine Kinase | at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kammerer RC, Di Stefano E, Schmitz D. A gas-liquid chromatography assay for phencyclidine and its metabolites. J Anal Toxicol. 1980 Nov-Dec;4(6):293-8. doi: 10.1093/jat/4.6.293. PMID 7206659
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12485966/